CLINICAL TRIAL: NCT04863378
Title: Efficacy of a Technology-Based Multimodal Brain Health Intervention for Older African Americans: The SHARP Study
Brief Title: Efficacy of a Multimodal Brain Health Intervention for Older African Americans
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Oregon Clinical and Translational Research Institute (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Raina Croff, Co-Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022363; KL2TR002370 (NIH)
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Impairment, Mild; Cognitive Decline
Keywords: social engagement; neighborhood walking; reminiscence; physical activity; African American; Mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive healthy participants (Experimental): Participants are Black/African American adults aged 65 or over who are cognitively healthy according to a baseline Montreal Cognitive Assessment score of 24 or higher. Participants continuously wear an actigraph watch to assess activity level. Daily sleep behavior is captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data is collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continue to wear the actigraph watch and continued to sleep on the sleep sensor, and walk 4-16 weeks with their triads. Triads walk 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) are accessed via the SHARP Walking Application via a group Android tablet device.
  Interventions: Behavioral: Walking conversational reminiscence
- Community stakeholder interviewees (No Intervention): Participants are Black/African American adults aged 55 and over who are individually interviewed to provide qualitative insight into salient historical landmarks and events to include in future walking routes for the Oakland area; Participants in this non-interventional group do not participate in study activities other than a qualitative interview.
- Mildly Cognitively Impaired (MCI) participants (Experimental): Participants are Black/African American adults aged 65 or over who are mildly cognitively impaired according to a baseline Montreal Cognitive Assessment score below 24. Participants continuously wear an actigraph watch to assess activity level. Daily sleep behavior is captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data is collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continue to wear the actigraph watch and continued to sleep on the sleep sensor, and walk 4-16 weeks with their triads. Triads walk 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) are accessed via the SHARP Walking Application via a group Android tablet device.
  Interventions: Behavioral: Walking conversational reminiscence

INTERVENTIONS:
Behavioral: Walking conversational reminiscence — Triadic walking with prompted conversational reminiscence
  Other Names: SHARP: Sharing History through Active Reminiscence and Photo-imagery
  Arms: Cognitive healthy participants; Mildly Cognitively Impaired (MCI) participants

SUMMARY:
This study tests the feasibility, acceptability, and efficacy of a multimodal intervention (walking, social engagement, and reminiscence), including the use of wearable digital biomarkers, for cognitively healthy and mildly cognitively impaired African Americans aged 65 and older.

DETAILED DESCRIPTION:
Cognitively healthy and mildly cognitively impaired participants engage in up to 8 weeks of baseline data collection and 4-16 weeks of triadic neighborhood walking using a group tablet device to access pre-programmed 1-mile routes. GPS (Global Positioning System)-triggered historical images of local Black culture and history along the route prompt conversational reminiscence about Portland, Oregon's historically Black neighborhoods. Digital biomarker technology (a continuously worn actigraph watch and an unobtrusive under-the-mattress sleep sensor) and weekly online surveys via a study Chromebook assess feasibility, acceptability, efficacy, and health outcomes. Intermittent discussions and check-ins with participants, and observational sessions will be used to elicit participant feedback.

ELIGIBILITY:
Inclusion Criteria for walkers:

1. Self-identified African American,
2. Age > 65 years old
3. Reside or resided for >10 years in Portland's historically Black neighborhoods (to be familiar with Memory Markers about this area),
4. Able to ambulate independently.
5. Meeting Cognition Criteria

   1. Participants with MCI (Mild Cognitive Impairment) will meet criteria consistent with the criteria outlined by the NIA-Alzheimer's Association workgroup
   2. Participants without cognitive impairment will have a Montreal Cognitive Assessment (MoCA) score > 24 (and not meet MCI criteria). Participants' cognitive function should allow them to get to and from walk locations independently or with minimal assistance.
6. Cognitive function allows independent (or minimally assisted) travel to and from walk locations
7. In-home reliable broadband internet (for weekly online surveys).
8. Ability to read, speak, and understand English

Exclusion Criteria:

1. Self-reported or clinically diagnosed dementia
2. Significant disease of the central nervous system
3. Severely depressed (CES-D score > 16), significantly symptomatic psychiatric disorder
4. Advanced cardiovascular disease that would make walking difficult, including history of congestive heart failure
5. Unstable insulin-dependent diabetes mellitus, received diagnosis Type 1 Diabetes, started insulin within past 3 months, hospitalized for hypoglycemia within past 6 months.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raina Croff, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Background] Croff RL, Witter Iv P, Walker ML, Francois E, Quinn C, Riley TC, Sharma NF, Kaye JA. Things Are Changing so Fast: Integrative Technology for Preserving Cognitive Health and Community History. Gerontologist. 2019 Jan 9;59(1):147-157. doi: 10.1093/geront/gny069. PMID 29961887

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants of the Community Stakeholder Interviewees group are identified via a consultation between the study team and representatives from UC Davis Alzheimer's Disease Center and the AAMLO
Groups:
- Cognitively Healthy Participants: Participants were Black/African American adults aged 65 or over who are cognitively healthy according to a baseline Montreal Cognitive Assessment score of 24 or higher. Participants continuously wore an actigraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
- Mildly Cognitively Impaired (MCI) Participants: Participants were Black/African American adults aged 65 or over who are mildly cognitively impaired according to a baseline Montreal Cognitive Assessment score below 24. Participants continuously wore an actigraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
- Community Stakeholder Interviewees: Participants were Black/African American adults aged 55 and over who were individually interviewed to provide qualitative insight into salient historical landmarks and events to include in future walking routes for the Oakland area
Period: Overall Study
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees
Started | 4 | 5 | 4
Completed | 4 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Community Stakeholder Interviewees: Participants were Black/African American adults aged 55 and over were individually interviewed to provide qualitative insight into salient historical landmarks and events to include in future walking routes for the Oakland area
- Total: Total of all reporting groups
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees | Total
Number analyzed (Participants) | 4 | 5 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 4 | 5 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (4.64) | 79.2 (4.36) | 66.5 (7.73) | 72.54 (4.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 13
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Daily Average Steps Recorded by Actigraphy Watch
Description: Daily steps are recorded on a continuously worn actigraphy watch (Withings), which measures 24-hour activity (gross motor activity).
Time Frame: 24 weeks
Population: Outcome measure data not collected from participants in the Community Stakeholder Interviewees group
Measure: Mean (Standard Deviation); unit: daily step count
Groups:
- Cognitively Healthy Walkers: Participants were Black/African American adults aged 65 or over who have healthy cognition. Participants continuously wore an ActiGraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
  Walking conversational reminiscence: Triadic walking with prompted conversational reminiscence
- Mildly Cognitively Impaired (MCI) Walkers: Participants were Black/African American adults aged 65 or over who are mildly cognitively impaired. Participants continuously wore an ActiGraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
Arm/Group | Cognitively Healthy Walkers | Mildly Cognitively Impaired (MCI) Walkers | Community Stakeholder Interviewees
Number analyzed (Participants) | 4 | 5 | 0
daily step count | 2570 (1000) | 1140 (1030) |

2. Primary Outcome: Daily Average Sleep Time Recorded by an Emfit QS Sleep Sensor
Description: Emfit QS under-the-mattress sleep sensor measured sleep-wake cycles per 24-hour period.
Time Frame: 24 weeks
Population: Outcome measure data not collected from participants in the Community Stakeholder Interviewees group
Measure: Mean (Standard Deviation); unit: hours of sleep per night
Arm/Group | Cognitively Healthy Walkers | Mildly Cognitively Impaired (MCI) Walkers | Community Stakeholder Interviewees
Number analyzed (Participants) | 4 | 5 | 0
hours of sleep per night | 6.71 (1.75) | 5.07 (1.84) |

3. Primary Outcome: Weekly Health Update Survey Response Time
Description: Participants completed a brief health update survey every week via their home computer or phone. Response time (the time it took each participant to complete the survey) was recorded in seconds.
Time Frame: 24 weeks
Population: Outcome measure data not collected from participants in the Community Stakeholder Interview group
Measure: Mean (Standard Deviation); unit: seconds to complete weekly survey
Groups:
- Cognitively Healthy Participants: Participants were Black/African American adults aged 65 or over who have healthy cognition. Participants continuously wore an actigraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
  Walking conversational reminiscence: Triadic walking with prompted conversational reminiscence
- Mildly Cognitively Impaired (MCI) Participants: Participants were Black/African American adults aged 65 or over who are mildly cognitively impaired. Participants continuously wore an actigraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees
Number analyzed (Participants) | 4 | 5 | 0
seconds to complete weekly survey | 195 (33.2) | 472 (234) |

4. Primary Outcome: Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire assessing sleep quality and sleep disturbances over a 1-month time period. The PQSI is composed of 19 query items, a combination of open-ended questions and Likert-type scales which are scored from 0 (no difficulty) to 3 (severe difficulty), and includes 7 sleep components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A global score is calculated from the sum of scores for each of the seven components. Total scores range from 0 to 21, a higher score indicates more acute sleep disturbances.
Time Frame: 24 weeks
Population: Outcome measure data not collected from participants in the Community stakeholder interviewees group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cognitively Healthy Participants: Participants were Black/African American adults aged 65 or over who have healthy cognition. Participants continuously wore an actigraph watch to assess activity level. Daily sleep behavior was captured on an under-the-mattress sleep sensor. Up to 8 weeks of baseline data was collected on participants prior to starting the walking component of the intervention. After the baseline data collection period, participants continued to wear the actigraph watch and continued to sleep on the sleep sensor, and walked 4-16 weeks with their triads. Triads walked 1-mile routes, three times a week while engaging in image-prompted conversational reminiscence recorded for a digital archive. Walking routes and GPS-linked reminiscence prompts (historical images with questions) were accessed via the SHARP Walking Application via a group Android tablet device.
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees
Number analyzed (Participants) | 4 | 5 | 0
score on a scale | 7.00 (4.55) | 5.60 (3.65) |

5. Primary Outcome: Weekly Survey Completion Rate
Description: Healthy and mildly cognitively impaired participants completed a weekly online health update survey, receiving weekly reminders to complete it. Survey completion rates and completion times over the study's duration is another measure of cognitive change.
Time Frame: 24 Weeks
Population: Outcome measure data not collected from participants in the Community Stakeholder Interviewees group
Measure: Number; unit: percentage of survey completion
Units Other Than Participants: surveys
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees
Number analyzed (Participants) | 4 | 5 | 0
Number analyzed (surveys) | 67 | 58 | 0
percentage of survey completion | 91 | 60 |

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Cognitively Healthy Participants: Participants were Black/African Americans aged 65 and over who are cognitively healthy according to a baseline Montreal Cognitive Assessment score of 24 or higher. Walkers continuously wear an actigraph watch to assess activity level. Daily sleep behavior is captured on an under-the-mattress sleep sensor. After up to 8 weeks of baseline data collection, participants walked 1-mile routes in triads, three times a week for 4-16 weeks while engaging in prompted conversational reminiscence recorded for a digital archive.
  Walking conversational reminiscence: Triadic walking with prompted conversational reminiscence
- Mildly Cognitively Impaired (MCI) Participants: Participants were Black/African Americans aged 65 and over who are mildly cognitively impaired according to a baseline Montreal Cognitive Assessment score below 24. Walkers continuously wear an actigraph watch to assess activity level. Daily sleep behavior is captured on an under-the-mattress sleep sensor. After up to 8 weeks of baseline data collection, participants walked 1-mile routes in triads, three times a week for 4-16 weeks while engaging in prompted conversational reminiscence recorded for a digital archive.
  Walking conversational reminiscence: Triadic walking with prompted conversational reminiscence
Arm/Group | Cognitively Healthy Participants | Mildly Cognitively Impaired (MCI) Participants | Community Stakeholder Interviewees
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT04863378/Prot_SAP_ICF_000.pdf